CLINICAL TRIAL: NCT03448302
Title: Computed Tomography Perfusion of Colorectal Cancer in Correlation With Tumor Grade
Brief Title: Computed Tomography Perfusion Colorectal Cancer With Tumor Grade
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Peter Edward Megala, Principal investigator, Assiut University
Other Study IDs: CTPCRCICWTG
Record Dates: First submitted 2018-02-22; First posted 2018-02-28 (Actual); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Colo-rectal Cancer
MeSH Terms: conditions — Colonic Neoplasms | interventions — Cytidine Triphosphate

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with colorectal adenocarcinoma: The patients will undergo computed tomography perfusion
  Interventions: Radiation: Computed tomography perfusion

INTERVENTIONS:
Radiation: Computed tomography perfusion — Pre-contrast images will be obtained to identify the colorectal tumor location. Then Fifty milliliters of iopromide (Ultravist ) will be injected intra-venously at rate of 5 milliliter per second via an automatic pump injector for computed tomography perfusion scans. Computed tomography perfusion scans will be performed at the mid-portion of the tumor for 60seconds beginning 5 seconds after contrast injection. Then arterial input will be defined by using the mouse to place a circular region of interest and the tumor region of interest will be placed on the most enhanced area of the tumor. Tumor blood flow, blood volume, mean transient time & permeability surface measurements will be obtained.

SUMMARY:
Colorectal cancer is the third most commonly diagnosed cancer in the world. The 5-years survival rate depends on the tumor stage and grade at patient presentation. Individual treatment strategy based on the tumor stage and grade should be applied to improve the prognosis, So the pre-operative diagnostic evaluation and grading of colorectal cancer are important.

DETAILED DESCRIPTION:
Diagnosis of cancer colon is usually based on colonoscopy which provides direct visualization of the lesions and allows for biopsies. However the pre-operative specimens from endoscopic biopsies sometimes fail to grade tumor because of the lack of sufficient tissue. Recent improvements in computed tomography have allowed for minimally invasive evaluation of cancer colon. Quantitative iodine density measurement can be used to differentiate low and high grade colorectal cancer. However, debate continues regarding the correlation between tumor grade and computed tomography perfusion parameters of colorectal cancer demonstrating the need for further investigation in this area of research.

ELIGIBILITY:
Inclusion Criteria:

* Any patient with primary colorectal mass

Exclusion Criteria:

* Colorectal mass pathologically proved to be benign Female patient at child bearing period with suspected pregnancy Raised renal chemistry Hypersensitivity to contrast.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with colorectal mass pathologically proved to be adenocarcinoma by colonoscpoic biopsy
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-03-10 (Estimated); Primary Completion 2019-03-10 (Estimated); Study Completion 2019-07-10 (Estimated)

PRIMARY OUTCOMES:
Blood flow of tumor | One month
  Accuracy of blood flow of the tumor in prediction of tumor grade in correlation with histopathological results

SECONDARY OUTCOMES:
Blood volume of the tumor | One month
  Accuracy of blood volume of the tumor in prediction of tumor grade in correlation with histopathological results
Mean transient time of the tumor | One month
  transient time of the tumor in prediction of tumor grade in correlation with histopathological results
Permeability surface of the tumor | One month
  Accuracy of permeability surface of the tumor in prediction of tumor grade in correlation with histopathological results

CONTACTS AND LOCATIONS:
Overall Officials: Peter E Megala, MBBCh, Principal Investigator — Assiut University
Locations (1):
- Faculty of Medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sun H, Xu Y, Yang Q, Wang W. Assessment of tumor grade and angiogenesis in colorectal cancer: whole-volume perfusion CT. Acad Radiol. 2014 Jun;21(6):750-7. doi: 10.1016/j.acra.2014.02.011. PMID 24809317
- [Background] Kim JW, Jeong YY, Chang NK, Heo SH, Shin SS, Lee JH, Hur YH, Kang HK. Perfusion CT in colorectal cancer: comparison of perfusion parameters with tumor grade and microvessel density. Korean J Radiol. 2012 Jan-Feb;13 Suppl 1(Suppl 1):S89-97. doi: 10.3348/kjr.2012.13.S1.S89. Epub 2012 Apr 23. PMID 22563293
- [Background] Goh V, Glynne-Jones R. Perfusion CT imaging of colorectal cancer. Br J Radiol. 2014 Feb;87(1034):20130811. doi: 10.1259/bjr.20130811. PMID 24434157
- [Background] Dighe S, Castellano E, Blake H, Jeyadevan N, Koh MU, Orten M, Swift I, Brown G. Perfusion CT to assess angiogenesis in colon cancer: technical limitations and practical challenges. Br J Radiol. 2012 Oct;85(1018):e814-25. doi: 10.1259/bjr/19855447. Epub 2012 Apr 18. PMID 22514101
- [Background] Marley AR, Nan H. Epidemiology of colorectal cancer. Int J Mol Epidemiol Genet. 2016 Sep 30;7(3):105-114. eCollection 2016. PMID 27766137